CLINICAL TRIAL: NCT03982732
Title: Maternal Antibody in Milk After Vaccination
Acronym: MAMA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: St George's, University of London (Other)
Collaborators: European Society for Paediatric Infectious Diseases (Other)
Responsible Party: Sponsor
Other Study IDs: 18.0068
Record Dates: First submitted 2019-06-10; First posted 2019-06-11 (Actual); Last update posted 2019-06-11 (Actual); Status verified 2019-06

CONDITIONS: Pertussis; Vaccination; Pregnancy; Breastmilk
MeSH Terms: conditions — Whooping Cough

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — We will collect samples of colostrum within the first 48 hours following delivery along with a blood sample and a further breastmilk sample at 2 and 6 weeks following delivery.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Women vaccinated at less than 24 weeks: Women receiving a pertussis containing vaccine at less than 24 weeks
  Interventions: Biological: Boostrix-IPV
- Women vaccinated at 24-27+6 weeks: Women receiving a pertussis containing vaccine at 24-27+6 weeks
  Interventions: Biological: Boostrix-IPV
- Women vaccinated at 28-31+6 weeks: Women receiving a pertussis containing vaccine at 28-31+6 weeks
  Interventions: Biological: Boostrix-IPV

INTERVENTIONS:
Biological: Boostrix-IPV — Receipt of Boostrix IPV at three different gestational time periods

SUMMARY:
Single-centre observational pilot study exploring pertussis specific antibody concentration in the breastmilk of women vaccinated against pertussis in pregnancy at different gestational ages. This study is made up of two stages: first stage to confirm recruitment methods and optimise the laboratory assay and a second stage to complete recruitment for the pilot study.

DETAILED DESCRIPTION:
Pertussis disease is a highly infectious respiratory illness caused by Bordetella pertussis, which can cause significant morbidity and mortality. There has been an increase in cases in many high income countries with high vaccination coverage and in an attempt to control this, antenatal vaccination programmes have been introduced in several countries, including the UK. Vaccination in pregnancy is a strategy which seeks to boost the maternal antibody levels, increase the placental transfer of antibody and consequently increase the antibody levels in the infant.

Human breast milk is a dynamic source of nutrition for the infant and is made up of many immunologically active components including antibody. The principal antibody in breastmilk is IgA and it has been shown that the amount of disease specific antibody in breastmilk can be increased by vaccination in pregnancy for a number of pathogens including pertussis. Secretory IgA (sIgA) plays an important role in immune exclusion in which it blocks adhesion of a pathogen onto a mucosal surface. As the first step of pertussis pathogenesis is the adhesion of bacteria to the ciliated respiratory epithelium in the nasopharynx and trachea there is a clear biological rationale for the hypothesis that receiving breast milk containing more IgA could enhance neonatal immunity and consequently the protective effects of vaccination in pregnancy.

The best time in pregnancy for administering the pertussis vaccination is debated in the literature, with some advocating vaccination in the second trimester and others supporting later vaccination to coincide the time of serum antibody peak with optimum placental transfer. This issue has been considered exclusively from the perspective of serum immunoglobulin G (IgG), but the impact of timing of vaccination in pregnancy on IgA levels in milk may also be important. Previous studies have shown that there is a peak in the pertussis specific IgA in breast milk at day 10 following vaccination, which then declines, and consequently there may be a significant difference in the amount of IgA available in the breastmilk for an infant born to a mother vaccinated at 20 weeks for example, compared to a mother vaccinated at 32 weeks. This may therefore have an impact on future guidelines on optimal time of vaccination in pregnancy.

ELIGIBILITY:
Inclusion Criteria:

* Singleton pregnancy
* Received pertussis vaccination between 16 and 32 gestational weeks
* Planning to breastfeed

Exclusion Criteria:

* Received vaccination outside of the 16-32 week window
* Not planning to breastfeed
* Diagnosis of an immunodeficiency syndrome
* Multiple pregnancy

Min Age: 18 Years | Sex: Female
Age Groups: Adult, Older Adult
Gender Based: Yes — Participant must have been vaccinated in pregnancy.
Study Population: Women who received a pertussis vaccination between 16 and 32 weeks and are pregnant or within 48 hours of delivery.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2018-08-07 (Actual); Primary Completion 2019-08-31 (Estimated); Study Completion 2019-10-31 (Estimated)

PRIMARY OUTCOMES:
Anti PT IgA at less than 48 hours in colostrum | Within 48 hours of delivery
  Anti-pertussis toxin (PT) Immunoglobulin A (IgA) concentration in colostrum

SECONDARY OUTCOMES:
Total IgA and IgG in colostrum and breastmilk | Within 48 hours and at 14 and 42 days after delivery
  Total IgA and IgG concentration in colostrum and breastmilk
Anti-PT IgA concentration in breastmilk | At 14 and 42 days following delivery
  Anti-PT IgA concentration in breastmilk
Anti-PT IgG concentration in colostrum and breastmilk | Within 48 hours and at 14 and 42 days after delivery
  Anti-PT IgG concentration in colostrum and breastmilk
Anti PT IgG concentration in maternal serum | Within 48 hours of delivery
  Anti PT IgG concentration in maternal serum

CONTACTS AND LOCATIONS:
Overall Officials: Kirsty Le Doare, Study Director — St George's, Univeristy of London
Locations (1):
- St Georges University Hospital NHS Foundation Trust, Tooting, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No